CLINICAL TRIAL: NCT02581683
Title: Does Magnesium Sulfate as a Supplement in Adductor Canal Blocks Improve Pain Control After Total Knee Arthroplasty?
Brief Title: Magnesium Sulfate in Adductor Canal Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Vidur Shyam, Assistant Professor, GFT, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAE-273-15
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Knee Arthroplasty
MeSH Terms: interventions — Magnesium Sulfate; Ropivacaine; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Magnesium (Experimental): Participants in this arm will receive magnesium sulfate + ropivacaine via adductor canal block
  Interventions: Drug: Magnesium Sulfate; Drug: Ropivacaine
- Non-magnesium (Active Comparator): Participants in this arm will receive ropivacaine via adductor canal block
  Interventions: Drug: Ropivacaine
- Sham (Sham Comparator): Participants in this arm will receive a sham adductor canal block
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Magnesium Sulfate — Given via adductor canal block
  Other Names: Sulfamag, Epsom salt, Health Canada DIN: 02139499
  Arms: Magnesium
Drug: Ropivacaine — Given via adductor canal block
  Other Names: Naropin
  Arms: Magnesium; Non-magnesium
Other: Sham — Sham adductor canal block
  Arms: Sham

SUMMARY:
Proper analgesia after total knee arthroplasty (TKA) is important for encouraging early ambulation, which can facilitate improved patient outcomes and early hospital discharge. For pain control after TKA, adductor canal blocks (ACBs) improve upon the gold standard femoral nerve blocks (FNBs) since they do not cause as much quadriceps muscle weakening, while providing equivalent analgesia. Multimodal analgesia has become commonplace as a method of superior pain control with fewer side effects. Magnesium sulfate as an adjuvant to FNB local anesthetics can improve pain control after surgery; however, it also prolongs time to ambulation. There are no reports on the effect of magnesium sulfate in ACBs on analgesia after TKA. Thus the purpose of this randomized, double-blind, controlled trial is to determine whether magnesium sulfate given with local anesthetics via ACB can prolong analgesia, reduce pain scores and opioid consumption, and increase mobilization in TKA patients.

DETAILED DESCRIPTION:
Adequate analgesia after surgery is important for patient well-being, satisfaction, rapid recovery, and timely discharge. Due to our aging population, total knee arthroplasties (TKAs) are an increasingly common surgical procedure in Canada, with 57,718 performed in 2012-2013 alone. Improved functional outcomes and early hospital discharge are facilitated when patients ambulate within several hours of surgery. Early ambulation is enabled by good analgesia without concomitant muscle weakness or debilitating side effects associated with opioid consumption. Given the high volume of knee replacements, the need to ambulate early, and the importance of effective pain management, the development of new analgesia techniques for TKAs is an important endeavor to reduce hospital costs and improve the quality of life of a substantial number of patients.

In order to minimize adverse side effects while still providing adequate postoperative analgesia, many anesthesiologists now co-administer smaller doses of several different medications, which act additively or synergistically depending on their combined and varied mechanisms of action. Often these medications are given locally, either directly into the knee (periarticularly) or near the nerves innervating the knee, for example the femoral nerve block (FNB) or the adductor canal block (ACB).

FNBs, wherein local anesthetic medications are injected around the femoral nerve, are commonly used to manage pain following TKA. Although they assist in providing quality postoperative pain relief, FNBs are also associated with weakening of the quadriceps muscle, and an increased risk of falls. The ACB involves an injection of local anesthetics such as ropivacaine or bupivacaine into the adductor canal in the middle third of the thigh, which contains the sensory saphenous nerve. ACB is as effective as FNB at reducing postoperative pain in TKA patients. However, ACBs do not cause quadriceps weakening to the same extent as FNBs, and result in earlier recovery of ambulation after surgery compared to FNBs. Since ACBs produce less quadriceps weakening (due to their actions on sensory, rather than motor, nerves), this anesthetic technique may reduce the risk of falling in the postoperative period compared to FNBs; however, most studies are underpowered to detect this statistically.

Recent attention has been given to magnesium sulfate (MgSO4) as a supplement to improve and/or prolong local anesthesia postoperatively. MgSO4 is thought to reduce pain via antagonism of N-methyl-D-aspartate (NMDA) receptors. A local mechanism of action on peripheral rather than central NMDA receptors is supported by studies showing that despite providing pain relief, peripherally administered MgSO4 does not increase cerebrospinal fluid concentrations of magnesium, implying that it cannot cross the blood-brain barrier to enter the central nervous system.

In knee surgery patients, locally administered MgSO4 via the periarticular route reduces postoperative pain, reduces cumulative analgesic consumption, and prolongs analgesia. MgSO4 co-administered with local anesthetic via FNB in knee surgery patients reduces pain and postoperative analgesic consumption compared to local anesthetic alone; however, it also prolongs the time to ambulation, which could delay hospital discharge. Currently, there are no investigations into the analgesic efficacy of MgSO4 administered via ACB in TKA patients. Therefore, the purpose of this randomized controlled trial is to assess the duration of analgesia in TKA patients receiving ACBs with or without MgSO4. The investigators hypothesize that patients receiving MgSO4 will have prolonged analgesia, improved pain scores, and will be able to mobilize further, all of which will contribute to a shorter hospital length of stay in these patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification score of 1 to 3
* Presenting for unilateral primary total knee arthroplasty
* age 18 to 85

Exclusion Criteria:

* inability to use a patient-controlled analgesia pump
* long-standing use of opioid medications (3 months or longer)
* history of chronic pain syndromes
* significant cardiovascular disease
* medical conditions that preclude the use of a regional anesthetic technique or any of the study drugs
* inability to read and understand English
* incompetent to give consent to study participation
* women who are pregnant or nursing

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic request | First occurrence during hospitalization (up to 72 hours postoperatively)
  Investigators will note the time lapsed between end of surgery and the first request for additional analgesia (given using patient controlled analgesia pumps, as is standard of care at the study institution).

SECONDARY OUTCOMES:
Cumulative morphine consumption | Cumulative dose during the first 24 postoperative hours
  Patient-controlled analgesia pumps allow the investigators to measure how much morphine each patient requests.
Number of steps taken | Number of steps taken during postoperative days 1 and 2
  The investigators will record the number of steps each patient takes during postoperative days 1 and 2 in hospital.
Pain | 2, 4, 8, 12, and 24 hours after adductor canal injection (or sham)
  Pain scores will be assessed using a visual analog scale at each of the above times.
Patient satisfaction | Once, 24 hours after surgery
  Patients will rate their satisfaction with their analgesia using a scale from 1 to 5.
Time to readiness for discharge | Once, upon occurrence, within 72 hours after surgery
  The time at which each patient reaches the criteria for discharge readiness determined by physiotherapy using an assessment checklist will be recorded.
Length of stay | Once, within 72 hours after surgery
  The length of hospital stay after surgery will be recorded for each patient
Side effects | Upon occurrence, up to 72 hours after surgery
  The incidence (presence/absence) of morphine-related side effects such as nausea, vomiting, itching, and respiratory depression will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Vidur Shyam, MBBS, FRCPC, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario

REFERENCES:
- [Background] Pavlin DJ, Rapp SE, Polissar NL, Malmgren JA, Koerschgen M, Keyes H. Factors affecting discharge time in adult outpatients. Anesth Analg. 1998 Oct;87(4):816-26. doi: 10.1097/00000539-199810000-00014. PMID 9768776
- [Background] Pavlin DJ, Chen C, Penaloza DA, Polissar NL, Buckley FP. Pain as a factor complicating recovery and discharge after ambulatory surgery. Anesth Analg. 2002 Sep;95(3):627-34, table of contents. doi: 10.1097/00000539-200209000-00025. PMID 12198050
- [Background] Jin F, Chung F. Multimodal analgesia for postoperative pain control. J Clin Anesth. 2001 Nov;13(7):524-39. doi: 10.1016/s0952-8180(01)00320-8. PMID 11704453
- [Background] Baratta JL, Gandhi K, Viscusi ER. Perioperative pain management for total knee arthroplasty. J Surg Orthop Adv. 2014 Spring;23(1):22-36. doi: 10.3113/jsoa.2014.0022. PMID 24641894
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Shah NA, Jain NP. Is continuous adductor canal block better than continuous femoral nerve block after total knee arthroplasty? Effect on ambulation ability, early functional recovery and pain control: a randomized controlled trial. J Arthroplasty. 2014 Nov;29(11):2224-9. doi: 10.1016/j.arth.2014.06.010. Epub 2014 Jun 19. PMID 25041873
- [Background] Jaeger P, Zaric D, Fomsgaard JS, Hilsted KL, Bjerregaard J, Gyrn J, Mathiesen O, Larsen TK, Dahl JB. Adductor canal block versus femoral nerve block for analgesia after total knee arthroplasty: a randomized, double-blind study. Reg Anesth Pain Med. 2013 Nov-Dec;38(6):526-32. doi: 10.1097/AAP.0000000000000015. PMID 24121608
- [Background] Mudumbai SC, Kim TE, Howard SK, Workman JJ, Giori N, Woolson S, Ganaway T, King R, Mariano ER. Continuous adductor canal blocks are superior to continuous femoral nerve blocks in promoting early ambulation after TKA. Clin Orthop Relat Res. 2014 May;472(5):1377-83. doi: 10.1007/s11999-013-3197-y. PMID 23897505
- [Background] Begon S, Pickering G, Eschalier A, Mazur A, Rayssiguier Y, Dubray C. Role of spinal NMDA receptors, protein kinase C and nitric oxide synthase in the hyperalgesia induced by magnesium deficiency in rats. Br J Pharmacol. 2001 Nov;134(6):1227-36. doi: 10.1038/sj.bjp.0704354. PMID 11704642
- [Background] Lysakowski C, Dumont L, Czarnetzki C, Tramer MR. Magnesium as an adjuvant to postoperative analgesia: a systematic review of randomized trials. Anesth Analg. 2007 Jun;104(6):1532-9, table of contents. doi: 10.1213/01.ane.0000261250.59984.cd. PMID 17513654
- [Background] Ko SH, Lim HR, Kim DC, Han YJ, Choe H, Song HS. Magnesium sulfate does not reduce postoperative analgesic requirements. Anesthesiology. 2001 Sep;95(3):640-6. doi: 10.1097/00000542-200109000-00016. PMID 11575536
- [Background] Mercieri M, De Blasi RA, Palmisani S, Forte S, Cardelli P, Romano R, Pinto G, Arcioni R. Changes in cerebrospinal fluid magnesium levels in patients undergoing spinal anaesthesia for hip arthroplasty: does intravenous infusion of magnesium sulphate make any difference? A prospective, randomized, controlled study. Br J Anaesth. 2012 Aug;109(2):208-15. doi: 10.1093/bja/aes146. Epub 2012 Jun 1. PMID 22661752
- [Background] Bondok RS, Abd El-Hady AM. Intra-articular magnesium is effective for postoperative analgesia in arthroscopic knee surgery. Br J Anaesth. 2006 Sep;97(3):389-92. doi: 10.1093/bja/ael176. Epub 2006 Jul 11. PMID 16835255
- [Background] Chen Y, Zhang Y, Zhu YL, Fu PL. Efficacy and safety of an intra-operative intra-articular magnesium/ropivacaine injection for pain control following total knee arthroplasty. J Int Med Res. 2012;40(5):2032-40. doi: 10.1177/030006051204000548. PMID 23206490
- [Background] Farouk S, Aly A. A comparison of intra-articular magnesium and/or morphine with bupivacaine for postoperative analgesia after arthroscopic knee surgery. J Anesth. 2009;23(4):508-12. doi: 10.1007/s00540-009-0822-8. Epub 2009 Nov 18. PMID 19921359
- [Background] Elsharnouby NM, Eid HE, Abou Elezz NF, Moharram AN. Intraarticular injection of magnesium sulphate and/or bupivacaine for postoperative analgesia after arthroscopic knee surgery. Anesth Analg. 2008 May;106(5):1548-52, table of contents. doi: 10.1213/ane.0b013e31816a67a8. PMID 18420874
- [Background] Ekmekci P, Bengisun ZK, Akan B, Kazbek BK, Ozkan KS, Suer AH. The effect of magnesium added to levobupivacaine for femoral nerve block on postoperative analgesia in patients undergoing ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2013 May;21(5):1119-24. doi: 10.1007/s00167-012-2093-4. Epub 2012 Jun 14. PMID 22696144
- [Background] Lee AR, Yi HW, Chung IS, Ko JS, Ahn HJ, Gwak MS, Choi DH, Choi SJ. Magnesium added to bupivacaine prolongs the duration of analgesia after interscalene nerve block. Can J Anaesth. 2012 Jan;59(1):21-7. doi: 10.1007/s12630-011-9604-5. Epub 2011 Oct 20. PMID 22012543
- [Derived] Zoratto D, Phelan R, Hopman WM, Wood GCA, Shyam V, DuMerton D, Shelley J, McQuaide S, Kanee L, Ho AM, McMullen M, Armstrong M, Mizubuti GB. Adductor canal block with or without added magnesium sulfate following total knee arthroplasty: a multi-arm randomized controlled trial. Can J Anaesth. 2021 Jul;68(7):1028-1037. doi: 10.1007/s12630-021-01985-5. Epub 2021 May 26. PMID 34041719